CLINICAL TRIAL: NCT01993420
Title: A Randomized, Double-blind, Vehicle Controlled Study of the Safety and Efficacy of Topical DRM02 in Subjects With Atopic Dermatitis
Brief Title: A Safety and Efficacy of DRM02 in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRM02-ADM02
Record Dates: First submitted 2013-11-15; First posted 2013-11-25 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DRM02 (Experimental): DRM02 Topical Gel, 0.25%
  Interventions: Drug: DRM02
- Vehicle (Placebo Comparator): DRM02 Topical Gel, Vehicle
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: DRM02
  Arms: DRM02
Other: Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine whether DRM02 is safe and effective in the treatment of atopic dermatitis when applied twice daily for 6 weeks.

DETAILED DESCRIPTION:
This is a double-blind, randomized, within-subject control, study enrolling 20 subjects with atopic dermatitis and designed to assess the safety, tolerability, and preliminary efficacy of DRM02.

Safety will be assessed during the study, through adverse events, local skin responses, urinalysis, serum chemistry and hematology laboratory testing, physical examination and vital signs.

Preliminary efficacy will be assessed through the Physician's Lesion Assessment (PLA) and the Eczema Area and Severity Index (EASI) from only the two lesions identified at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 70 years of age.
* Clinical diagnosis of stable atopic dermatitis (AD) and with two lesions of similar size and have an identical score of at least 5 but no more than 9 on the sum of the individual components of the Eczema Area and Severity Index (EASI) at the Target Lesion scale.
* Male or non-pregnant, non-lactating females.
* Signed informed consent.

Exclusion Criteria:

* Subjects who have unstable atopic dermatitis (AD).
* Significant infection at the target lesion site.
* Prior or concomitant use of systemic therapies for AD within the past 4 weeks. - Prior or concomitant use of topical treatments for AD, to within 10 cm of the target lesion within the past 4 weeks.
* Prior or concomitant use of oral retinoids for AD within the last 6 months.
* Use of biologics for AD within the past 3 months, or 5 half-lives (whichever is longer).
* Subjects who have poor skin condition within 5 cm of the target lesion.
* Subjects who are current drug or alcohol abusers; have a history of immunodeficiency disease; or are a poor medical risk because of other systemic diseases or active uncontrolled infections.
* Subjects with an unstable medical condition or a medical condition not adequately controlled with standard medical therapy.
* Subjects who are actively participating in an experimental therapy study or who have received experimental therapy within 30 days.
* Subjects who have a clinically significant laboratory value at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in Physician's Lesion Assessment | Week 6

SECONDARY OUTCOMES:
Physician's Lesion Assessment analyzed for treatment effect | From baseline to weeks 1, 2, 3, 4 and 6

OTHER OUTCOMES:
Physician's Lesion Assessment dichotomized into "success" and "failure" | Week 6
Severity of Target Lesion EASI scores | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Beth Zib, Study Director — Dermira, Inc.
Locations (2):
- Canada (2):
  - Clinique Médicale Dr Isabelle Delorme, Drummondville, Quebec
  - Innovaderm Research, Inc, Montreal, Quebec